CLINICAL TRIAL: NCT03521362
Title: MyT1DHero: A Randomized Controlled Trial of an mHealth Intervention to Improve Parent-child Communication and Adolescent Self-management of Type 1 Diabetes
Brief Title: MyT1DHero: an mHealth Intervention for Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Corewell Health West (Other); American Diabetes Association (Other)
Responsible Party: Principal Investigator, Bree Holtz, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MyT1DHeroRCT
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type1diabetes
Keywords: mHealth; Adolescent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyT1DHero App (Experimental): Participants in this group will receive use of the MyT1DHero app.
  Interventions: Device: MyT1DHero
- "Other" T1D App (Active Comparator): Participants in this group will receive use of a different app with less capabilities.
  Interventions: Device: Other T1D Mobile App

INTERVENTIONS:
Device: MyT1DHero — MyT1DHero is an app with two separate interfaces, one for the parent and one for the child, that work together to help them communicate about diabetes management. The child receives system reminders to enter their blood glucose numbers, and parents receive a notification about each blood glucose test their child enters. Parents are also able to use the app to communicate with their child about their plan for care. The app has customizable blood glucose reminders and ranges, videos of support from other adolescents with T1D, snack lists, and other educational information on T1D.
  Arms: MyT1DHero App
Device: Other T1D Mobile App — A mobile app will be used in this control/comparison group that only has blood sugar testing reminders and logging capabilities. There will be no other components of the app.
  Arms: "Other" T1D App

SUMMARY:
The overall objective of the proposed research is to improve HbA1c, adherence to treatment plans, and family communication surrounding adolescents' self-management of T1D. The investigators will test the efficacy of the MyT1DHero app against an attention control group. This will allow investigators to better understand the health and psychosocial improvements being made through the app.

DETAILED DESCRIPTION:
This research seeks to realize the potential and test the efficacy of MyT1DHero to improve adolescent users' glycemic control and adherence to blood glucose monitoring. The investigators' goal is to help families receive more social support, and to improve diabetes knowledge, self-efficacy, family communication, and quality of life. The investigators further seek to decrease family conflict among children with T1D and their parents. In a 12-month RCT, investigators will randomize 166 adolescents and their parents to one of two groups: (1) attention control, or (2) the MyT1DHero app. Adolescents enrolled in the study will be 10-15 years old, and will have been living with T1D for <1 year or >5 years at the start of the study. The primary outcome will be a change in the participants' HbA1C from baseline levels at the start of the study, to levels measured after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The adolescents must:

  1. have a T1D diagnosis according to the ADA practice guidelines,
  2. be 10 to 15 years old,
  3. have had a diagnosis of T1D for at least six months,
  4. have an HbA1c > 7,
  5. have had at least two outpatient visits in the past two years,
  6. be treated at Spectrum for diabetes,
  7. be fluent in English,
  8. have a parent/guardian willing to participate,
  9. have and be allowed to use a mobile phone for the study, and
  10. have permission from their care team to participate.

The parent/guardian must:

1. have an adolescent with T1D who is 10 to 15 years old,
2. be fluent in English, and
3. have daily access to email and the Internet (for appointment reminders and technical support).

Exclusion Criteria:

* For the adolescents include:

  1. significant medical conditions other than T1D,
  2. being treated for thyroid disorders, celiac disease, or eating disorders, and
  3. being in foster care.

Exclusion criteria for both the adolescents and parents/guardians include:

(a) a diagnosis of a major psychiatric or neurocognitive disorder (e.g., traumatic brain injury, dementia, schizophrenia, bipolar disorder, borderline personality disorder, and intellectual and developmental disabilities.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Diabetes Behavior Rating Scale at 12 months | Baseline and 12 months
  A measure of diabetes adherence for both parent and child participants. Never (1) - Always(5) with a higher score indicating better adherence.
Change from Baseline HbA1c at 6 months and 12 months | Baseline, 6 months, and 12 months
  A laboratory test that measures how high blood glucose has been on average over the last 8-12 weeks - for child participants only (Lower number is best)

SECONDARY OUTCOMES:
Change from Baseline PROMIS Item Bank v2.0 - Informational Support - Short Form 6a at 12 months | Baseline and 12 months
  A measure of social support for the parent participants. Never (1) - Always (5), with a higher score indicating better support.
Change from Baseline PROMIS Item Bank v2.0 - Emotional Support - Short Form 8a at 12 months | Baseline and 12 months
  A measure of social support for the parent participants. Never (1) - Always (5), with a higher score indicating more support.
Change from Baseline NIH Toolbox Emotional Support (Ages 8-17) at 12 months | Baseline and 12 months
  A measure of social support for the child participants. Never (1) - Always (5), with a higher score indicating more support.
Change from Baseline Diabetes Empowerment Scale Short Form at 12 months | Baseline and 12 months
  A measure of diabetes-related self-efficacy for both parent and child participants. Strongly disagree (1) - Strongly agree (5), with a higher score indicating more empowerment.
Change from Baseline PROMIS® Item Bank v.1.0 - General Self-Efficacy at 12 months | Baseline and 12 months
  A measure of self-efficacy for the parent participants. I am not at all confident (1) - I am very confident (5), with a higher score indicating higher self-efficacy.
Change from Baseline NIH Toolbox Self-efficacy (ages 8-12) at 12 months | Baseline and 12 months
  A measure of self-efficacy for the child participants. Never (1) - Very often (5), with a higher score indicating higher self-efficacy.
Change from Baseline Confidence in Diabetes Self-Care (Psychometric properties of a new measure of diabetes-specific self-efficacy in Dutch and U.S. patients with type 1 diabetes) at 12 months | Baseline and 12 months
  A measure of diabetes-related self-efficacy for the child participants. Strongly disagree (1) - Strongly agree (5), with a higher score indicating more confidence in self-care ability.
Change from Baseline PROMIS® Item Bank v1.0 - General Life Satisfaction - Short Form 5a at 12 months | Baseline and 12 months
  A measure of quality of life for the parent participants. Strongly disagree (1) - Strongly agree (7), with a higher score indicating more life satisfaction.
Change from Baseline PedsQL (Measurement Model for the Pediatric Quality of Life Inventory) at 12 months | Baseline and 12 months
  A measure of quality of life for the child participants. Never (0) - Almost Always (4), with a lower score indicating better quality of life.
Change from Baseline Neuro-QOL Item Bank v1.0 -Pediatric Stigma - Short Form at 12 months | Baseline and 12 months
  A measure of stigma for the child participants. Never (1) - Always (5), with a higher score indicating more feelings of stigma.
Change from Baseline Diabetes Conflict Scale at 12 months | Baseline and 12 months
  A measure of conflict for both the parent and child participants. Almost Always (1) - Never (3), with a higher score indicating less conflict.
Change from Baseline PROMIS® Parent Proxy Item Bank v1.0 - Family Relationships - Short Form 8a at 12 months | Baseline and 12 months
  A measure of family characteristics for both the parent and child participants. Never (1) - Always (4), with a higher score indicating better family relationships.
Change from Baseline Diabetes Family Behavior Scale at 12 months | Baseline and 12 months
  A measure of family characteristics for both the parent and child participants. All of the time (1) - Never (5), with a lower score indicating better family behavior.
Change from Baseline Family Functioning Scale at 12 months | Baseline and 12 months
  A measure of family characteristics for both the parent and child participants. Totally disagree (1) - Totally agree (6). Responses are summed. Subscales include intimacy (items 1, 4, 6, 10, 13, 15, 18, 20, 23, 26, 27, 29), conflict (items 3, 5, 8, 9, 12, 14, 17, 19, 22, 24), and parenting style (items 2, 7, 11, 16, 21, 25, 28, 30).
Change from Baseline Impact on Family (Construct: Parental perceptions of the impact of a child's medical condition on the family) at 12 months | Baseline and 12 months
  A measure of family characteristics for the parent participants. Strongly disagree (1) - Strongly agree (5), with a higher score indicating more impact (burden).
Change from Baseline Family Satisfaction (FSS) at 12 months | Baseline and 12 months
  A measure of family characteristics for the parent participants. Very dissatisfied (1) - Extremely satisfied (5), with a higher score indicating more satisfaction.
Change from Baseline Neuro-QOL Item Bank v1.0 -Anxiety - Short Form at 12 months | Baseline and 12 months
  A measure of anxiety for the parent participants. Never (1) - Always (5), with a higher score indicating more anxiety.
Change from Baseline Neuro-QOL Item Bank v1.0 -Pediatric Anxiety - Short Form at 12 months | Baseline and 12 months
  A measure of anxiety for the child participants. Never (1) - Almost always (5), with a higher score indicating more anxiety; Not at all (1) - Very much (5); with a higher score indicating more anxiety.
Change from Baseline Short-Form Outcome Expectations at 12 months | Baseline and 12 months
  A measure of diabetes outcome expectancy for both the parent and child participants. Strongly disagree (1) - Strongly agree (5), with a higher score indicating more positive outcome expectations
Usability and Satisfaction Questionnaire | 12 months
  A measure of technology usability and satisfaction for both the parent and child participants
Unified theory of acceptance and use of technology (UTAUT) Vantakesh, Morris, et al., 2003 | 12 months
  A measure of technology usability and satisfaction for both the parent and child participants

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study Website — http://myt1d.org/wordpress/